CLINICAL TRIAL: NCT03215004
Title: Developing a Functional Cure for HIV Disease: Clinical Specimen Collection From HIV Positive Individuals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: American Gene Technologies International Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AGT-CS168
Record Dates: First submitted 2017-07-07; First posted 2017-07-12 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: HIV Infections
Keywords: Volunteer; HIV; Leukapheresis
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — HIV positive samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical specimens are required from HIV positive individuals with viremia controlled by antiretroviral therapy to complete process development for a genetically modified autologous T cell product, AGT103-T. The product will be used in a subsequent early stage clinical trial in subjects with chronic HIV disease and viremia suppressed by antiretroviral therapy as the initial step in testing a functional cure for HIV disease. Enrolled participants provide a venous blood specimen (approximately 25mL) to determine their level of HIV-reactive CD4+ T cells. Subjects with positive T cell responses will be asked to undergo leukapheresis and their clinical specimens will be used to validate and qualify the AGT103-T cell product.

DETAILED DESCRIPTION:
This protocol is to collect blood specimens from HIV positive individuals. The first blood draw will be done at the first study visit and if eligible, the second blood collection will be done via leukapheresis at the second visit. The leukapheresis procedures will follow the facility's standard operating procedures and protocol requirements for leukapheresis.

Volunteers will be males or females between and including the ages of 18 years and 60 years. Volunteers will provide written informed consent and meet all inclusion and exclusion criteria. Each participant can be in the study for up to 120 days (3 months).

The study will be conducted in accordance with GCP/ICH for human research for the purposes of obtaining clinical specimens for research. There is no endpoint for this study, however, data collected from this study will include, but not be limited to, gender, demographics, medical history, clinical laboratory values, and volume of the blood collected. The data will be summarized in future studies reporting results from a planned clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between ≥18 and ≤60 years
* Documented HIV infection for at least 3 years prior to study entry
* Stable on HIV antiretroviral regimen with viral suppression to <50c/mL plasma for >2 years
* Agrees not to change antiretroviral regimen (unless medically indicated) during the study period
* CD4+ T cell count >500 cell per millimeter cubed (cells/mm3) at last measurement within 6 months of study participation
* CD4+ T cell nadir of >350 cells/mm3
* HIV plasma viral load <50 copies of viral RNA per milliliter (mL) for >2 years
* Participants who had intermittent, isolated episodes of detectable low-level viremia (<500c/mL; blips) will remain eligible.
* Have not received cytoreduction therapy within 3 months of study entry
* Do not have prior events of hemorrhagic cystitis
* Is not being treated or does not have bacteremia within the past 6 months
* Does not have signs or symptoms of acute infectious disease
* Adequate venous access and no other contraindications for leukapheresis
* Hematocrit is >33% or hemoglobin is ≥13g/dL (males) and ≥12g/dL (females) at last measurement within 7 days prior to study enrollment; test also required within 3 days prior to leukapheresis
* Weighs more than 75 lbs
* Not pregnant at time of enrollment
* Ability to understand the study and must be willing to comply with study-required procedures and visits, including only changing antiretroviral regimen when indicated by the study doctor during the study period
* Written informed consent signed and dated by study participant

Exclusion Criteria:

* Acute or chronic hepatitis B or hepatitis C infection with detectable viremia
* Any viral hepatitis or liver disease (e.g. cirrhosis)
* Active or recent (prior 6 months) AIDS defining complication
* Any experimental HIV medications within the past 12 weeks
* Cancer or malignancy that has not been in remission for at least 5 years with the exception of successfully treated basal cell carcinoma of the skin
* Current diagnosis of NYHA grade 3 or 4 congestive heart failure or uncontrolled angina or arrhythmias
* Any clinically significant renal, hepatic, and pulmonary disease
* Inadequate venous access or contraindicated for leukapheresis
* Significant laboratory values and/or a chronic medical condition that, in the opinion of the Principal Investigator, could impact trial participation
* Receiving another investigational drug or device within 30 days of study entry
* Previously received any gene transfer therapy
* History or any features on physical examination indicative of a bleeding diathesis
* Use of chronic corticosteroids, hydroxyurea, or immunomodulating agents (e.g. interleukin-2, interferon-alpha or gamma, granulocyte colony stimulating factors, etc.) within 30 days prior to screening (NOTE: Use of inhaled or topical steroids is not exclusionary)
* Breast-feeding or pregnant
* Use of aspirin, dipyridamole, warfarin or any other medication that is likely to affect platelet function or other aspects of blood coagulation during the 2-week period prior to leukapheresis
* Active drug or alcohol use or dependence that, in the opinion of the Investigator, would interfere with adherence to study requirements
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to study entry
* Recent vaccination or intercurrent illness within 5 weeks prior to T cell infusion (NOTE: It is recommended that participants should have completed their routine vaccinations, e.g. hepatitis A or B, pneumococcus, influenza and tetanus diphtheria booster, at least 30 days prior to screening for the study)
* Asplenia: any conditions resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema or idiopathic angioedema

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals with chronic, persistent HIV disease that is well-controlled by combination antiretroviral therapy
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2017-07-25 (Actual); Primary Completion 2021-02-07 (Estimated); Study Completion 2021-02-07 (Estimated)

PRIMARY OUTCOMES:
Collection of clinical specimens | up to 120 days
  The blood samples collected will be tested to measure the absolute and relative levels of CD4+ and CD8+ T cells. Data will describe the range of CD4+ T cell and CD8+ T cell responses to peptide stimulation. The samples will also help validate the assays and processes for the development of the cell product to be used in a future clinical trial.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Providence Hospital, Washington D.C., District of Columbia
  - Institute of Human Virology, University of Maryland Baltimore, Baltimore, Maryland